CLINICAL TRIAL: NCT00100503
Title: Cortical Reorganization Following Pediatric Constraint-Induced Therapy
Brief Title: Brain Reorganization Following Constraint-Induced Therapy in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050066; 05-N-0066
Record Dates: First submitted 2004-12-31; First posted 2005-01-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-08-30

CONDITIONS: Cerebral Palsy
Keywords: Rehabilitation; Forced Use; Hemiplegia; Magnetic Resonance Imaging; TMS; Cerebral Palsy; Spastic Hemiplegia; Healthy Volunteer; HV
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

SUMMARY:
This study will examine how therapy changes the way the brain controls movements in children with cerebral palsy. Normally, one side of the brain controls movements in the opposite side of the body. In cerebral palsy, however, this pattern may be different, with one side of the brain controlling movements on the same side of the body. This study will use magnetic resonance imaging (MRI) and transcranial magnetic stimulation (TMS) to study brain function in children with cerebral palsy before and after therapy.

Children between 9 and 17 years of age with spastic hemiplegia type cerebral palsy will be recruited for this study from the National Rehabilitation Hospital and Georgetown University Center Medical Center in Washington, D.C., and the Sparks Center at UAB in Alabama. In addition, five healthy control children will be recruited from community groups, such as Cub Scouts, Brownies, and schools. Candidates are screened with a review of medical records and neurological and physical examinations.

Healthy controls undergo MRI (described below) twice, 3 weeks apart. Children with cerebral palsy undergo the following tests and procedures:

1. Rehabilitation evaluation at the NIH Clinical Center Rehabilitation Medicine Department.
2. MRI: For this test, the child lies on a table that slides in and out of the MRI scanner-a metal cylinder surrounded by a strong magnetic field. He or she wears earplugs to muffle loud knocking sounds that occur during scanning. Images are obtained while the child performs simple finger tapping movements.
3. Movement Testing:

   1. Finger tapping: The child taps buttons on a box hooked up to a computer
   2. Muscle reflex measurements: One method uses a small motor that makes the child's fingers move with sudden, small movements; a second method uses small shocks to the finger or wrist. The shocks feel like a buzz; most are gentle, but some might feel stronger.
4. TMS: This procedure maps brain function. A wire coil is held on the scalp, and a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. During the stimulation, the child may be asked to perform simple movements.. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the child may hear a click and feel a pulling sensation on the skin under the coil.
5. Therapy: After these tests, children are randomly selected to receive either standard therapy (neurodevelopmental treatment) or constraint-induced therapy, as follows:

   1. Neurodevelopmental therapy uses principles of movement science to enhance the child's capacity to function. The child receives therapy a few times a week for 3 weeks.
   2. Constraint-induced therapy uses a combination of motor learning method and constraint to teach the new motor skills in the child's affected hand. Children treated with this therapy must live near a special treatment center in Alabama for the 3 weeks of treatment. The child's good arm is constrained with a bivalve, removable cast. The cast is placed before therapy starts and remains in place except when the therapist removes it once a day to examine the good arm. With the cast on, children are encouraged to use their affected hand in new ways. The therapist then uses the motor learning method, building motor programs as a result of practice, to teach them new skills. Motor learning therapy is 6 hours a day.
6. Post-treatment testing: After treatment, children undergo repeat rehabilitation assessment, MRI, TMS, and movement testing.

DETAILED DESCRIPTION:
Objective: To determine the underlying brain reorganization that occurs in children with hemiplegic cerebral palsy before and after pediatric Constraint-Induced therapy.

Background: A promising new therapy for adults with hemiparesis consequent to stroke, known as Constraint-Induced Movement (CI) therapy, has recently been modified for use in children with cerebral palsy. Children with cerebral palsy treated with CI therapy show significant gains in motor skills after receiving this intensive and extended treatment.

There is evidence to suggest that, after an acute stroke in adults, the undamaged motor cortex exerts greater control over movements in the affected hand than is normally seen in neurologically intact subjects. While this might seem to be an advantage, combined functional magnetic resonance imaging (fMRI) and transcranial magnetic stimulation (TMS) studies demonstrate that it is associated with poor motor recovery in adults after a stroke and impaired hand function in patients with cerebral palsy. Thus, anomalous motor control of the affected hand by the unaffected cortex may reflect a less efficient cortical reorganization process.

There is controversy about how CI therapy produces an improvement in motor function. Conflicting evidence from fMRI and TMS studies in adult patients with stroke have shown that patients may have either an increase in ipsilateral motor cortical activation or an increase in activation in the damaged hemisphere. The answer to this controversy may be related to the presence of ipsilateral projections. Since ipsilateral projections are associated with worse functional outcome, determining the type of response to CI therapy may give insights into those patients who need more intense therapy.

Subject Population: Children with hemiplegic subtype of cerebral palsy; age-matched children with no neurological abnormalities

Design: We will assess motor cortex activation before and after CI therapy using fMRI and neurophysiologic tests including TMS and muscle reflex studies in children with hemiplegic cerebral palsy with and without evidence for ipsilateral projections.

Outcome measures: Patients will be stratified by the presence of mirror movements. Primary outcome measure will be laterality index on cortical activation of the fMRI before and after CI therapy. Secondary outcome measures will be standardized measures of sensory and motor function. We will examine the relationship between the presence of anomalous ipsilateral motor control and cortical reorganization following CI therapy.

Significance: Understanding this relationship is essential for planning large randomized controlled trials. Since anomalous ipsilateral cortical reorganization reflects an inefficient cortical reorganization process, treatment outcome of CI therapy may also be worse in this group. In this case, future studies may need to stratify children on study entry according to types of brain reorganization.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Children 9 to 17 years of age.

     Cerebral palsy patients:
  2. Children previously diagnosed with spastic hemiplegia subtype of cerebral palsy
  3. Children with non-progressive cerebral lesions acquired pre-, peri- or post-natally, before 1 year of age.

Typically Developing subjects:

1. Scores below 60 on Connor's attention deficit/hyperactivity disorder (ADHD) checklist.
2. Normal neurological history and examination

EXCLUSION CRITERIA:

1. Any child who is pregnant
2. Patients with Development Quotient (DQ) or Intelligence Quotient (IQ) below 50 on standardized tests

   Cerebral palsy patients:
3. Children with subtypes of cerebral palsy that are not hemiplegia.
4. Children with uncontrolled seizures within the last 6 months
5. Children with progressive or neurodegenerative disorders; underlying known genetic or chromosomal disorders, familial or non-familial syndromes (without known chromosomal or genetic defect)
6. Patients with cerebral lesions caused by sickle cell disease or by emboli associated with congenital cardiac lesions
7. Patients incapable of voluntary movement or with severe cognitive deficits who cannot follow simple verbal commands

Typically Developing Children:

1. Children with chronic medical disorders or any neurological and /or psychiatric disorder including attention deficit hyperactivity disorder or learning disorder
2. Children taking regular medications, including medications for allergies, hormonal oral contraceptives, or over-the-counter medications
3. Children born before 36 weeks gestation as estimated by dates, ultrasound or other methods (if a discrepancy exists, then the ultrasound estimation will be taken as definitive)

Exclusionary criteria for clinical MRI studies:

1. Any child with metal objects in the body such as pacemakers, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses, cochlear implants, or shrapnel fragments).
2. Any child with permanent tattoos on the eyelids (ferromagnetic iron oxide-based) tattoo pigments can interact with the static magnetic field of an MRI imager.

Exclusionary criteria for TMS:

1. Children with hearing loss (greater than 15 dB at any individual frequency) in either ear (as evaluated in the Audiology Department, CC, NIH).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50
Dates: Start 2004-12-27; Study Completion 2006-08-30

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Carr LJ, Harrison LM, Evans AL, Stephens JA. Patterns of central motor reorganization in hemiplegic cerebral palsy. Brain. 1993 Oct;116 ( Pt 5):1223-47. doi: 10.1093/brain/116.5.1223. PMID 8221056